CLINICAL TRIAL: NCT00002809
Title: Unrelated Bone Marrow Transplantation With Cyclophosphamide and Total Body Irradiation For Hematologic Malignancies and Bone Marrow Failure States
Brief Title: Bone Marrow Transplant Plus Cyclophosphamide and Total-Body Irradiation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Temple University Bone Marrow Transplant Program, Temple University Health Systems
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064937; TUHSC-2803; NCI-V96-0950
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; refractory anemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; secondary acute myeloid leukemia; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Antilymphocyte Serum; Filgrastim; sargramostim; gamma-Globulins; Cyclophosphamide; Methotrexate; Tacrolimus; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: sargramostim
Biological: therapeutic immune globulin
Drug: cyclophosphamide
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy and radiation therapy together with bone marrow transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bone marrow transplant from an unrelated donor together with cyclophosphamide and total-body irradiation works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Study the curative potential of high-dose cyclophosphamide and total-body irradiation followed by rescue with bone marrow from volunteer HLA-matched donors in patients with a variety of hematologic malignancies and bone marrow failure states.
* Study the toxic effects associated with matched unrelated bone marrow transplantation in this patient population.
* Participate in collaborative research studies with the National Marrow Donor Program.

OUTLINE: All patients receive myeloablative therapy with high-dose cyclophosphamide and total body irradiation over 4 days; patients with severe aplastic anemia also receive antithymocyte globulin. Patients then undergo allogeneic bone marrow transplantation. Filgrastim (G-CSF) is given after transplant to accelerate engraftment. Sargramostim (GM-CSF) may be given in case of graft failure.

All patients receive graft-versus-host-disease (GVHD) prophylaxis with tacrolimus, methotrexate, and gamma globulin. Established GVHD is treated with corticosteroids and, as necessary, antithymocyte globulin.

Patients are followed at 100 days, 6 months, and 1 year after transplant, then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients per year will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following hematologic malignancies/disorders:

  * Acute lymphoblastic leukemia

    * In second or subsequent complete remission (CR)
    * In first CR with high-risk features (e.g., Philadelphia chromosome-positive)
    * In first relapse and failed conventional salvage therapy
  * Acute myelogenous leukemia (AML)

    * In second or subsequent CR
    * In early first relapse
    * In full first relapse and failed conventional salvage therapy
    * In first CR with high-risk features, e.g., trisomy 8 or FAB 6/7

      * Standard-risk AML offered conventional-dose consolidation chemotherapy or autologous bone marrow transplantation
  * Chronic myelogenous leukemia in chronic, accelerated, or second chronic phase

    * No blast crisis
  * Severe aplastic anemia that has failed at least 1 course of immunosuppressive therapy
  * Paroxysmal nocturnal hemoglobinuria with high-risk features (e.g., disseminated intravascular coagulation, thrombotic events)
  * Myelodysplastic syndrome, i.e.:

    * Symptomatic, transfusion-dependent refractory anemia with excess blasts
    * (RAEB) or RAEB in transformation
  * Secondary leukemia in CR following conventional-dose induction chemotherapy
* Unrelated marrow donor available who is 8 out of 10-, 9 out of 10-, or 10 out of 10-antigen serologically HLA-matched at A, B, C, DRb, and DQB loci by molecular typing
* No CNS malignancy

PATIENT CHARACTERISTICS:

Age:

* 17 to 60

Performance status:

* Karnofsky 70-100%

Life expectancy:

* No reduction due to other serious illness

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 3 mg/dL
* AST/ALT no greater than twice normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Left ventricular ejection fraction at least 45%
* No severe hypertension

Pulmonary:

* DLCO, FEV_1, and FVC at least 50%

Other:

* HIV negative
* No active infection at time of transplant
* No advanced diabetes
* No significant neurologic deficit
* No active drug or substance abuse
* No emotional disorders
* Able to participate in frequent medical care for at least 1-2 years
* Willing to comply with National Marrow Donor Program policies

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 1996-08; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth F. Mangan, MD, FACP, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania, United States